CLINICAL TRIAL: NCT04685954
Title: Clinical Comparison of Bulk-fill and Incremental Composite Resin Restorations
Brief Title: Clinical Comparison of Bulk-fill and Incremental Composite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dr. Fatma Dilşad Öz, Assoc. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bulk-incremental
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-12

CONDITIONS: Tooth Disease
MeSH Terms: conditions — Tooth Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bulk-Fill (Experimental): Filtek™ Bulk Fill Posterior, 3M ESPE, St. Paul MN, USA (FB)
  Interventions: Device: Filtek Bulk-Fill Posterior
- Incremental (Experimental): Filtek Ultimate Universal, 3M ESPE, St. Paul MN, USA (FU)
  Interventions: Device: Filtek Ultimate Universal

INTERVENTIONS:
Device: Filtek Bulk-Fill Posterior — Bulk-fill restorative composite
  Arms: Bulk-Fill
Device: Filtek Ultimate Universal — Incremental restorative composite
  Arms: Incremental

SUMMARY:
The clinical performance of a 5-mm bulk-fill and an incremental resin composite in class II restorations will be evaluated and compared. After recruiting participants with at least 2 approximal caries lesions, all restorations will be placed by a single clinician. All caries lesions will be removed before restoring. Cavities will be divided into two groups: a 5 mm bulk-fill composite resin [Filtek™ Bulk Fill Posterior, 3M ESPE, St. Paul MN, USA (FB)] and an incremental posterior composite resin [Filtek Ultimate Universal, 3M ESPE, St. Paul MN, USA (FU)] All restorative procedures will be conducted according to manufacturers' instructions. Restorations will be scored using modified United States Public Health Service (USPHS) criteria after a week (baseline) 6, 12, 24, 36 and 48 months. Descriptive statistics will be performed using chi-square tests.

ELIGIBILITY:
Inclusion Criteria:

* age range will be 18 to 65
* patients should have at least 2 approximal caries lesions require restoration
* healthy periodontal status
* a good likelihood of recall availability

Exclusion Criteria:

* poor gingival health
* adverse medical history
* potential behavioral problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performances of different restorative systems according to USPHS criteria | two years
  Two year results according to USPHS criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No